CLINICAL TRIAL: NCT01852006
Title: Abdominal Binding: a Novel Intervention to Relieve Dyspnea and Improve Exercise Tolerance in Patients With Chronic Obstructive Pulmonary Disease?
Brief Title: Abdominal Binding in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Dennis Jensen, Ph.D., Assistant Professor, McGill University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RI MUHC 3234
Record Dates: First submitted 2013-05-07; First posted 2013-05-13 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- COPD AB ON (Experimental): Abdominal Binder "ON"
  Interventions: Device: Abdominal Binder
- COPD AB OFF (No Intervention): Abdominal Binder "OFF" (control)

INTERVENTIONS:
Device: Abdominal Binder — Abdominal Binding to increase end-expiratory gastric pressure by 5-8 centimetres of water at rest.
  Other Names: McDavid Inc., 493R Universal Back Support
  Arms: COPD AB ON

SUMMARY:
Conventional approaches to relieve dyspnea (respiratory discomfort) in chronic obstructive pulmonary disease (COPD) have focused on improving respiratory motor drive (e.g., hyperoxia) and/or dynamic respiratory mechanics (e.g., bronchodilators). Although these approaches yield meaningful symptom improvements there remains many COPD patients incapacitated by dyspnea. Accumulating evidence suggests that abdominal binding (AB) is a potentially novel method of improving respiratory muscle function and, by extension, dyspnea and exercise tolerance in COPD. Thus, the purpose of this randomized, cross-over study is to test the hypothesis that AB improves exertional dyspnea and exercise tolerance in symptomatic patients with COPD by improving dynamic respiratory muscle function. To this end, the investigators will examine the effects of AB on detailed assessments of baseline pulmonary function (spirometry, plethysmography), dyspnea (sensory intensity & affective responses), neural respiratory drive (diaphragm EMG), contractile respiratory muscle function (esophageal, gastric & transdiaphragmatic pressures), ventilation, breathing pattern and cardiometabolic function during symptom-limited constant load cycle exercise (75% Wmax) in 20 patients with GOLD stage II/III COPD.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Aged ≥40 years
* Ambulatory
* Cigarette smoking history ≥15 pack years
* No change in medication dosage or frequency of administration, with no exacerbations or hospitalization in the preceding 6 weeks.
* Post-bronchodilator Forced Expiratory Volume in 1 second between 30-80% predicted
* Post-bronchodilator Forced Expiratory Volume in 1 second/forced vital capacity ratio of <70%

Exclusion Criteria:

* Presence of active cardiopulmonary disease other than COPD
* Use of domiciliary oxygen
* Exercise-induced arterial blood oxyhemoglobin desaturation to <80% on room air.
* Body Mass Index <18.5 or ≥35 kg/m2.
* Allergy to latex
* Allergy to lidocaine or its "caine" derivates.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Sensory Intensity (Borg 0-10 scale) ratings of dyspnea at isotime during exercise | Patients will be followed until all study visits are complete, an expected average of 2 weeks

SECONDARY OUTCOMES:
Exercise Endurance Time (EET) | Patients will be followed until all study visits are complete, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Jensen, Ph.D., Principal Investigator — McGill University
Locations (1):
- Montreal Chest Institute; McGill University Health Center & McGill University, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Abdallah SJ, Smith BM, Wilkinson-Maitland C, Li PZ, Bourbeau J, Jensen D. Effect of Abdominal Binding on Diaphragmatic Neuromuscular Efficiency, Exertional Breathlessness, and Exercise Endurance in Chronic Obstructive Pulmonary Disease. Front Physiol. 2018 Nov 14;9:1618. doi: 10.3389/fphys.2018.01618. eCollection 2018. PMID 30487757
- See also: Clinical Exercise & Respiratory Physiology Laboratory (CERPL) of McGill University — http://www.mcgill.ca/cerpl